CLINICAL TRIAL: NCT06385925
Title: Phase 1/2 Study of TSN1611 in Subjects With Advanced Solid Tumors Harboring KRAS G12D Mutation
Brief Title: A Study of TSN1611 Treating Patients With Advanced Solid Tumors Harboring KRAS G12D Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tyligand Pharmaceuticals (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSN1611-2023-101
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasm
Keywords: solid tumor; KRAS G12D mutation; pancreatic cancer; colorectal cancer; non-small cell lung cancer; malignant neoplasm
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Taxes; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Dose-finding/evaluation of TSN1611 monotherapy (Experimental): The phase 1 part will evaluate the prespecified sequential dose levels of TSN1611 in subjects with KRAS G12D mutant advanced solid tumors to determine the recommended dose of TSN1611 for further investigation.
  Interventions: Drug: TSN1611
- Phase 2: Dose expansion of TSN1611 monotherapy (Experimental): Phase 2 part will evaluate the efficacy and safety of TSN1611 as monotherapy at the recommended dose level in separate groups of patients with pancreatic cancer, colorectal cancer, non-small cell lung cancer, or other solid tumors, harboring KRAS G12D mutations.
  Interventions: Drug: TSN1611
- Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort A (Experimental): Cohort A: TSN1611 combined with cetuximab treating subjects with advanced solid tumors harboring KRAS G12D mutation:
  Interventions: Drug: TSN1611
- Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort B (Experimental): Cohort B: TSN1611 combined with GnP regimen (i.e., gemcitabine and nab-paclitaxel) treating subjects with advanced PDAC with KRAS G12D mutation who received no prior systemic treatment in the advanced setting.
  Interventions: Drug: TSN1611
- Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort C (Experimental): Cohort A3: subjects with advanced NSCLC harboring KRAS G12D mutation who received no more than three prior systemic treatment regimens in the advanced setting.
  Interventions: Drug: TSN1611

INTERVENTIONS:
Drug: TSN1611 — TSN1611 will be administered at the assigned dose level, orally, until disease progression or intolerable toxicity.
  Arms: Phase 1: Dose-finding/evaluation of TSN1611 monotherapy; Phase 2: Dose expansion of TSN1611 monotherapy
Drug: TSN1611 — TSN1611 BID, Cetuximab will be administered via intravenous infusion at a dose of 500 mg/m² every 2 weeks.
  Arms: Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort A
Drug: TSN1611 — TSN1611 BID, Paclitaxel (albumin-bound) at 125 mg/m² and gemcitabine at 1000 mg/m² will be administered via intravenous infusion on Days 1, 8, and 15 of each 4-week cycle.
  Other Names: Paclitaxel (albumin-bound)
  Arms: Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort B
Drug: TSN1611 — TSN1611 BID everyday and Patients will be administered with mFOLFOX6 on Days 1 and 2, every 2 weeks.
  Other Names: Oxaliplatin injection; fluorouracil; leucovorin
  Arms: Dose of Phase 1b/2 part of TSN1611 combination therapy-Cohort C

SUMMARY:
The study is a first-in-human (FIH), open-label, multi-center phase 1/2 study of TSN1611 in subjects with KRAS G12D mutant advanced solid tumors. This study will consist of a phase 1 dose escalation part and phase 2 dose expansion part. This study will evaluate the efficacy of TSN1611 at RP2D(s) through ORR using RECIST version 1.1, and determine and confirm the MTD/RP2D for TSN1611 in combination with cetuximab, in combination with cetuximab and mFOLFOX6, in combination with gemcitabine and albumin-bound paclitaxel in subjects with selected solid tumors.

DETAILED DESCRIPTION:
Phase 1 Part of TSN1611 Monotherapy:

The phase 1 part will evaluate the prespecified dose levels of TSN1611. Dose escalation will continue until up to the highest planned dose or the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is determined. Dose optimization could be performed as indicated by the emerging data.

Phase 2 Part of TSN1611 Monotherapy:

hase 2 part of TSN1611 monotherapy will evaluate the efficacy and safety of TSN1611 as monotherapy at the RP2D until disease progression or unacceptable toxicity in separate groups of patients with pancreatic cancer, colorectal cancer, non-small cell lung cancer, or other solid tumors, harboring KRAS G12D mutations.

Phase 1b/2 Part of TSN1611 Combination Therapy:

This part will consist of the investigations of 3 combined therapies (Cohort A, B and C). In each cohort, there will be a Phase 1b Safety Lead-in Stage to determine the dose of TSN1611 for the combination therapy (this part will be conducted in selected sites), followed by the Phase 2 Expansion Stage to enroll more subjects to determine the efficacy in different cohorts.

ELIGIBILITY:
Subjects must meet all the following inclusion criteria to be eligible for participation in this study:

* The subject fully understands the requirements of the study and voluntarily signs the ICF.
* At least 18 years of age at the time of informed consent.≤ 75 years of age for Cohort B and C.
* Life expectancy of 3 months or more.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Phase 1 part (1a/1b) of Monotherapy:

Subjects with histologically or cytologically confirmed locally advanced or metastatic solid tumor harboring KRAS G12D mutation; subjects must be refractory or intolerable to standard treatment, or have no standard treatment available, or the subject is ineligible or declines standard treatment.

Phase 2 part of TSN1611 Monotherapy:

Subjects with histologically or cytologically confirmed locally advanced or metastatic PDAC、CRC and NSCLC harboring KRAS G12D mutation; According to the requirements of different combined cohorts, the number of previous treatments is taken into account.

• Patients with adequate cardiac, liver, renal function, etc.

Exclusion Criteria

Subjects will be excluded if they meet any of the following criteria:

* Leptomeningeal disease or Active central nervous system (CNS) metastases.
* Prior systemic anti-cancer treatment within 21 days or 5 half-lives (whichever is shorter will be used as the criteria) prior to the first dose of study drug.
* Radical radiation within 4 weeks prior to the first dose of study drug; palliative radiotherapy within 1 week prior to the first dose of study drug.
* Any unresolved Grade 2 or higher toxicity from previous anticancer therapy except alopecia.
* Has participated in a study of investigational agent and received the investigational agent within 21 days or 5 half-lives, if known (whichever is shorter) prior to the first dose of study drug.
* History of interstitial lung disease (ILD), drug induced IDL, or current active pneumonitis, radiation pneumonitis requiring therapeutic intervention, or uncontrolled other lung disease.
* Any of the following in the past 6 months: myocardial infarction, unstable angina, symptomatic congestive heart failure, stroke or transient ischemic attack, pulmonary embolism.
* Prior treatment with KRAS G12D targeted therapy.
* Has a history or current evidence of any severe condition, concurrent therapy, or laboratory abnormality that might confound the interpretation of the study results, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) in phase 1 part | 21 days
  To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose(s) (RP2D[s]) of TSN1611 as monotherapy in subjects with KRAS G12D mutant advanced solid tumors.
Objective response rate (ORR) in phase 2 part | Up to 3 years
  To evaluate the anti-tumor activity of TSN1611 using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Adverse events | Up to 3 years
  To assess the safety profile and tolerability of TSN1611 as monotherapy in subjects with KRAS G12D mutant advanced solid tumors.
Area under the plasma concentration-time curve (AUC) | 9 weeks
  To characterize the pharmacokinetic (PK) profile of TSN1611.
Maximum blood concentrations (Cmax) | 9 weeks
  To characterize the PK profile of TSN1611.
Time to maximum blood concentration (Tmax) | 9 weeks
  To characterize the PK profile of TSN1611.
Duration of response (DOR) | Up to 3 years
  To evaluate the anti-tumor activity of TSN1611 using RECIST version 1.1.
Time to response (TTR) | Up to 3 years
  To evaluate the anti-tumor activity of TSN1611 using RECIST version 1.1.
Disease control rate (DCR) | Up to 3 years
  To evaluate the anti-tumor activity of TSN1611 using RECIST version 1.1.
Progression free survival (PFS) | Up to 3 years
  To evaluate the anti-tumor activity of TSN1611 using RECIST version 1.1.
Overall survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Li, Study Director — Tyligand Bioscience (Shanghai) Limited
Locations (19):
- United States (3):
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- China (16):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University - Donghu District, Nanchang, Jiang
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital - Zhejiang University School of Med, Hangzhou, Zhejiang
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Beijing Cancer Hospital, Beijing, China, Beijing
  - Shanghai Chest Hospital, Shanghai, China, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai, China, Shanghai

IPD SHARING:
Plan to Share IPD: No